CLINICAL TRIAL: NCT02590393
Title: The Role of Nicotine and Non-Nicotine Alkaloids in E-Cigarette Use and Dependence
Acronym: Ecig1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00059780; 1R01DA038554-01 (NIH)
Record Dates: First submitted 2015-10-27; First posted 2015-10-29 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking; E-cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nicotine + NNTAs (Experimental): Participants will be asked to switch from cigarette use to use of e-cigarettes for eight weeks. E-cigarette cartridges will contain tobacco extract with nicotine + NNTAs in a vehicle of propylene glycol and vegtable glycerin, with tobacco or menthol flavor matched to each participant's preference. The yields of nicotine and NNTAs will be in the range of typical commercial cigarettes.
  Interventions: Combination Product: E-cigarettes

INTERVENTIONS:
Combination Product: E-cigarettes — Participants will be asked to switch from cigarette use to use of e-cigarettes for eight weeks.
  Other Names: Electronic Nicotine Delivery System (ENDS); e-cigs; electronic cigarettes

SUMMARY:
The advent of electronic cigarette (e-cigarette) technologies represents one of the most significant developments in the last several decades, and provides a novel and promising strategy for substantially reducing the morbidity and mortality associated with smoking. However, serious concerns have been raised regarding the possibility that e-cigarettes will sustain a dependency on nicotine and that they may lead to continued use of conventional cigarettes known to be extremely harmful to health. Cigarette addiction critically involves a dependence on nicotine, but it is likely that other tobacco constituents contribute to dependence as well. Recent evidence suggests that non-nicotine tobacco alkaloids, or NNTAs (including anabasine, anatabine, nornicotine, and myosmine) may play a role in tobacco dependence. These alkaloids have been shown to augment the reinforcing effects of nicotine in animal models and to affect cravings in human smokers. E-cigarettes contain variable quantities of nicotine and NNTAs, but there is virtually no information available concerning the role of e-cigarette nicotine or NNTA content in influencing the concurrent use of cigarettes and e-cigarettes, when smokers attempt to switch from conventional combustible cigarettes to e-cigarettes. Additionally, it is not known whether the presence of nicotine and NNTAs in e- cigarettes may sustain dependence, making it difficult to relinquish these products. The proposed project will assess the acceptability, extent of switching behavior, and degree of dependence maintained when smokers are provided with e-cigarettes containing nicotine and NNTAs.

DETAILED DESCRIPTION:
A single group of thirty smokers will be recruited for the study to provide initial data to inform follow-up randomized controlled trials.

Dependence and concurrent use of e-cigarettes and cigarettes will be assessed by a battery of self-report, biochemical, and behavioral indices. This is not a tobacco cessation study and there is no intent to use e-cigarettes as a smoking cessation treatment. Smokers will be asked to use the e-cigarettes instead of their regular cigarettes during the study. E-cigarettes will not be used for the purpose of reducing urges, withdrawal or nicotine dependence; and e-cigarettes will not be described or used as a medical device or therapy.

Specific Aim 1: To assess the extent of switching from combustible cigarettes to e-cigarettes delivering nicotine along with NNTAs.

Switching will be assessed by self-report diaries and by reductions in expired air carbon monoxide, an index of combustible cigarette use.

Specific Aim 2: To assess the acceptability of e-cigarettes delivering nicotine along with NNTAs.

Ratings of user satisfaction and other subjective effects will be collected from participants, for both their customary brand of cigarettes and the e-cigarette to be used.

Specific Aim 3: To determine the extent of dependence maintained during use of e-cigarettes delivering nicotine with NNTAs, as well as the relationship between dependence and self-reported use of cigarettes and e-cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Have no known serious medical conditions;
* Are 21-65 years old;
* Smoke an average of at least 10 cigarettes per day;
* Have smoked at least one cumulative year;
* Have an expired air CO reading of at least 10ppm;
* Are able to read and understand English.

Potential subjects must agree to use acceptable contraception during their participation in this study. Potential subjects must agree to avoid the following during their participation in this study:

* Participation in any other nicotine-related modification strategy outside of this protocol;
* Use of tobacco products other than cigarettes, including pipe tobacco, cigars, snuff, and chewing tobacco;
* Use of e-cigarettes other than the ones provided during the study;
* Use of experimental (investigational) drugs or devices;
* Use of illegal drugs.

Exclusion Criteria:

* Actively seeking treatment for nicotine dependence;
* Uncontrolled high blood pressure (self-report);
* Coronary heart disease with symptoms (e.g., chest pain);
* Heart attack in the past year;
* Cardiac rhythm disorder (irregular heart rhythm with symptoms);
* Chest pain in the last month (unless history indicates a non-cardiac source);
* Symptomatic heart disorder such as heart failure;
* Advanced liver or kidney disease that requires medication or dialysis, paracentesis;
* Bleeding stomach ulcers in the past 30 days;
* Lung disease that requires oxygen;
* Major brain disorder (including stroke with residual deficit, brain tumor, and seizure disorder);
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Diabetes with insulin use;
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition (as determined by study medical provider);
* Diagnosis of thought disorder; such as bipolar disorder or schizophrenia;
* Psychiatric hospitalization within the past 12 months;
* Pregnant or nursing mothers;
* Use (within the past 7 days) of illegal drugs (or if the urine drug screen is positive for THC, Cocaine, Amphetamine, Opiates, Methamphetamines, PCP, Benzodiazepines, or Barbiturates), unless recent use of prescription opiates or benzodiazepines were taken for management of acute symptoms (e.g., tooth extraction, recent surgery, or sleep);
* Use of experimental (investigational) drugs within the past 7 days;
* Use of psychiatric medications including antidepressants and anti-psychotics may be permitted if the condition is stable (study medical provider discretion).
* Use of opiates, benzodiazepines, and muscle relaxants (unless taken for sleep or acute symptoms such as tooth extraction or recent surgery) within the past 7 days (study medical provider discretion);
* Use of Wellbutrin, bupropion, Zyban, Chantix, varenicline, nicotine patch, nicotine replacement therapy, clonidine or any other smoking cessation aid within the past 30 days;
* Use of cigars, pipes, Hookah, dissolvable nicotine, snuff, chewing tobacco, or e-cigarettes within the past 7 days;
* Diagnosis of alcohol abuse or dependence or self-report of consuming more than 6 drinks on one occasion more than one day per week;
* Significant adverse reaction to nicotine patch in the past;
* Current or recent participation (in the past 30 days) in another smoking treatment study at our Center or another research facility;

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

PRIMARY OUTCOMES:
Change in expired air carbon monoxide (CO) to assess recent smoking | Weeks 1-8
  Self-reported changes in cigarette use from baseline to week 8, expressed as a percentage of baseline values, will be calculated, based on expired air carbon monoxide readings.

SECONDARY OUTCOMES:
Mean volume of e-cigarette solution used per day to assess e-cigarette use. | Weeks 1-8
  The mean volume of solution used per day (by measuring the content and number of pods returned) will be calculated for each week.
Change in cigarette use, assessed by self-report in daily dairies | Weeks 1-8
  Self-reported changes in cigarette use from baseline to week 8, expressed as a percentage of baseline values, will be calculated, based on cigarette consumption recorded in daily diaries.
E-cigarette use, assessed by self-report in daily dairies | Weeks 1-8
  The self-reported use of e-cigarette pods, based on daily diaries, will be totaled for each week.
Change in Nicotine dependence | Weeks 1-8.
  The change in level of nicotine dependence will be assessed by administering the Fagerstrom Test for Nicotine Dependence questionnaire, administered at baseline and at week 8.
Satisfaction ratings | Weeks 1-8.
  The satisfaction of the experimental e-cigarette formulation will be assessed using the modified Cigarette Evaluation Questionnaire, with wording adapted to e-cigarettes.

CONTACTS AND LOCATIONS:
Overall Officials: Jed Rose, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke Center for Smoking Cessation, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No